CLINICAL TRIAL: NCT05176912
Title: Effects of Reformer Pilates Exercise Training in Overweight and Obese Women
Brief Title: Effects of Reformer Pilates Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Özge Gökalp, Principal Investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/02
Record Dates: First submitted 2021-12-03; First posted 2022-01-04 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Physical Performance
Keywords: Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Exercise Group (Experimental): Reformer Pilates exercises will given for 8 weeks, 3 days in a week.
  Interventions: Other: Exercise
- Control Group (No Intervention): Nothing given to the control group, will be told to continue their normal life for 8 weeks.

INTERVENTIONS:
Other: Exercise — Reformer Pilates exercises will given for 8 weeks, 3 days in a week
  Arms: Experimental Exercise Group

SUMMARY:
Aim: The aim of the study is to investigate the effects of Reformer Pilates exercises in overweight and obese woman.

Method: 47 sedentary overweight and obese women aged 30-60 years will be included in the study. Subjects will be divided into two groups: Reformer Pilates and control. The exercise group will be given Reformer Pilates training session 3 times a week over an 8-weeks period. Before and after the study, the subjects will be test for body composition with the bioelectrical impedance and for upper limb strength with the hand grip dynamometer. Moreover, the strength of the back muscle will be measure with the back dynamometer and the strength of the abdominal muscle with the sit-up test. Furthermore, the endurance of trunk, abdominal and back muscles will be measure with the McGill endurance tests. The endurance of the lower limb will be measure with the 30 second sit and stand test, and the balance with the Fullerton Advanced Balance Scale. Finally, the sleep quality will be measure with the Pittsburgh Sleep Quality Index, and the anxiety with the Hospital Anxiety and Depression Scale.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer female individuals between the ages of 30-60 years,
* BMI: 25 kg/m² and above,
* Individuals who have not surgery in the last 6 months,
* Individuals who have a medical report stating that there is no obstacle in terms of health,
* Individuals whose physical activity level will be determined by the International Physical Activity Questionnaire (IPAQ) will be included in the study.

Exclusion Criteria:

* Individuals with any neurological, orthopedis, cardiovascular, psychological problems,
* Individuals with any systemic disease (DM, cancer),
* Individuals who doing regular physical activity/sport in the last 6 months.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Change in the body composition to be evaluated by a bioelectrical impedance | Baseline and at the end of 8 weeks.
  fat mass and fat-free mass will be evaluated

SECONDARY OUTCOMES:
Change in the level of upper extremity strength to be evaluated by a hand grip dynamometer. | Baseline and at the end of 8 weeks.
  The subject sits upright in a supported chair and on a flat surface. The person is prepared with the knee and hip in 90⁰ flexion, forearm in neutral position and wrist in 0-30⁰ extension. During the measurement, the person whose grip strength is measured is asked to squeeze the arms of the dynamometer strongly.

OTHER OUTCOMES:
Change in the level of trunk flexor muscle endurance to be evaluated by a McGill core endurance tests. | Baseline and at the end of 8 weeks.
  The trunk flexor endurance test begins with the person in a sit-up position with the back resting against a jig angled at 60 degrees from the floor. Both knees and hips are flexed 90 degrees, the arms are folded across the chest with the hands placed on the opposite shoulder, and the feet are secured. After the apparatus is removed, the person maintains the isometric posture for as long as possible.
Change in the level of back extensors muscle endurance to be evaluated by a McGill core endurance tests. | Baseline and at the end of 8 weeks.
  The back extensors are tested with the upper body cantilevered out over the end of the test bench and with the pelvis, knees, and hips secured. The upper limbs are held across the chest with the hands resting on the opposite shoulders.
Change in the level of lateral muscle endurance to be evaluated by a McGill core endurance tests. | Baseline and at the end of 8 weeks.
  The lateral muscle is tested with the person lying in the full side-bridge position.
Change in the strength of the back to be evaluated by back dynamometer. | Baseline and at the end of 8 weeks.
  Back dynamometer: The measure strength of back muscles. Subject stand with knees fully extended and head and back straight. They use over-under grip with the bar across the thighs. They should pull the bar straight up by rolling shoulders without bending them back.
Change in the strength of the abdominal muscle to be evaluated by sit-up test. | Baseline and at the end of 8 weeks.
  Sit-up test: The measure strength of abdominal muscles. The subjects lying on the floor supine position. The knees are flexed at an angle of 90°, and an assistant supports the ankles. The subject raises upper body and then returns to the starting position.
Change in the endurance of the lower extremity to be evaluated by 30 second sit and stand test. | Baseline and at the end of 8 weeks.
  The chair-stand test administer using a folding chair without arms, with a seat height of 17 inches (43.2 cm). The test begin with the participant seated in the middle of the chair, back straight, feet approximately shoulder-width apart and placed on the floor at an angle slightly back from the knees. Arms cross at the wrists and held against the chest. At the signal 'go', the participant rise to a full stand and then return back to the seated position. The participants encourage to complete as many full stands as possible within 30-s time limit.
Change in the balance to be evaluated by Fullerton Advanced Balance Scale. | Baseline and at the end of 8 weeks.
  The Fullerton Test is mainly intended to identify highly-active older adults who are at an increased risk to experience fall-related injuries due to sensory impairments. The test uses both dynamic and static balance under different situations to identify balance deficits in older adults.
Change in the sleep quality to be evaluated by Pittsburgh Sleep Quality Index. | Baseline and at the end of 8 weeks.
  The Pittsburgh Sleep Quality Index, a self-administered questionnaire, includes four open-ended questions and 14 questions to be answered using event-frequency and semantic scales. The tool looks at seven areas; subjective sleep quality, sleep latency (the time it takes to fall asleep), sleep duration, habitual sleep efficiency (the ratio of total sleep time to time in bed), sleep disturbances, the use of sleep-promoting medication, and daytime dysfunction.
Change in the anxiety level to be evaluated by Hospital Anxiety and Depression Scale (HADS) . | Baseline and at the end of 8 weeks.
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measureanxiety and depression (7 items for each subscale). Thetotal score is the sum of the 14 items, and for each sub-scale the score is the sum of the respective seven items(ranging from 0-21).

CONTACTS AND LOCATIONS:
Overall Officials: Berkiye Kirmizigil, Asst. Prof, Study Chair — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gokalp O, Kirmizigil B. Effects of reformer pilates on body composition, strength, and psychosomatic factors in overweight and obese women A randomized controlled trial. Sci Rep. 2025 Jul 2;15(1):23602. doi: 10.1038/s41598-025-09683-8. PMID 40603682